CLINICAL TRIAL: NCT06424587
Title: The Effect of Music Intervention on Anxiety, Fear, and Pain in Pediatric Patients Receiving Intrathecal Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Hatice Uzşen, Research assistant, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IT
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Nurse's Role
Keywords: anxiety; hematology-oncology nursing; pain intervention; randomized controlled trial; fear
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: a parallel group, randomized, controlled experimental study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music intervention group (Experimental): In addition to the routine practice of the clinic, the pediatric patients in this group listened to music through headphones for 20 minutes just before the procedure to reduce the child's anxiety and fear. The therapeutic effect of music was used. Before the study, children between the ages of 6 and 12 who were inpatients at the clinic were asked what music they most liked to listen to, what kind of music they liked, and what their favorite artists and songs were. The music was selected based on the children's answers. In addition, the researcher added children's songs by a musician named Banu Kanıbelli.
  Interventions: Behavioral: Music intervention
- Control Group (No Intervention): Children were verbally informed about the treatment process and invasive procedures from the day they were diagnosed with the disease. The children in this group were verbally informed by the nurse in charge of the clinic about the intrathecal chemotherapy treatment and why it was performed

INTERVENTIONS:
Behavioral: Music intervention — : In addition to the routine practice of the clinic, the pediatric patients in this group listened to music through headphones for 20 minutes just before the procedure to reduce the child's anxiety and fear. The therapeutic effect of music was used. Before the study, children between the ages of 6 and 12 who were inpatients at the clinic were asked what music they most liked to listen to, what kind of music they liked, and what their favorite artists and songs were. The music was selected based on the children's answers. In addition, the researcher added children's songs by a musician named Banu Kanıbelli
  Arms: Music intervention group

SUMMARY:
Intrathecal chemotherapy is often used to prevent the spread of cancer to the central nervous system in pediatric patients and is one of the most invasive procedures. It is believed that the way it is administered and the complications experienced after treatment negatively affect the comfort of the pediatric patient, leading them to refuse the treatment.

DETAILED DESCRIPTION:
Receiving sedation is one of the pharmacological procedures for intrathecal chemotherapy which creates a particularly difficult situation for the child. However, since pharmacological methods increase the cost and cause toxicity in children, in recent years, the symptoms that occur in cancer treatment have been tried to be controlled with non-pharmacological methods. Music intervention facilitates a sense of control in patients and provides mental distraction, emotional smoothness, and relaxation, which have been found to have pain relief effects.

ELIGIBILITY:
Inclusion Criteria:

* To be between 6-12 years old,
* Being treated in the Hematology and Oncology Clinic,
* About to receive intrathecal chemotherapy treatment,
* The child not having pain before intrathecal chemotherapy treatment

Exclusion criteria were,

* Refusing to participate in the study,
* Being under 6 years of age and over 10 years of age,
* The child having pain prior to intrathecal chemotherapy treatment,
* Having any physical or mental disability,
* Not being able to speak Turkish.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
anxiety | 30 minutes before intrathecal chemotherapy treatment and just after music intervention
  Child Anxiety Meter-State (CAM-S):The scale can be scored between 1 and 10. An increase in the score means an increase in anxiety.
fear | 30 minutes before intrathecal chemotherapy treatment and just after music intervention
  Children's Fear Scale (CFS): The scale can be scored between 0 and 4. An increase in the score means an increase in fear
pain scale | 60 minutes after intrathecal chemotherapy treatment
  Face, Legs, Activity, Cry, Consolability pain scale (FLACC): total score between 0 and 10 is obtained by assigning 0, 1, or 2 points for each category. As the severity of pain increases, the total score increases, and as the severity of pain decreases,

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Uzsen, PhD, Principal Investigator — ondokuz mayıs üniversity
Locations (1):
- Ondokuz Mayis University, Samsun, Black Sea, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No